CLINICAL TRIAL: NCT01941199
Title: A Randomized, Open-label, Multiple Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of DA-1229 5 mg and Metformin IR 1000 mg After Oral Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of DA-1229 and Metformin After Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA1229_DIM_I
Record Dates: First submitted 2013-09-09; First posted 2013-09-13 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Metformin

ARMS (6):
- D → M → D+M (Experimental): D : DA-1229 5mg qd, M : metformin 1000mg bid
  Interventions: Drug: DA-1229; Drug: metformin; Drug: DA-1229 + metformin
- D → D+M → M (Experimental): D : DA-1229 5mg qd, M : metformin 1000mg bid
  Interventions: Drug: DA-1229; Drug: metformin; Drug: DA-1229 + metformin
- M → D → D+M (Experimental): D : DA-1229 5mg qd, M : metformin 1000mg bid
  Interventions: Drug: DA-1229; Drug: metformin; Drug: DA-1229 + metformin
- M → D+M → D (Experimental): D : DA-1229 5mg qd, M : metformin 1000mg bid
  Interventions: Drug: DA-1229; Drug: metformin; Drug: DA-1229 + metformin
- D+M → M → D (Experimental): D : DA-1229 5mg qd, M : metformin 1000mg bid
  Interventions: Drug: DA-1229; Drug: metformin; Drug: DA-1229 + metformin
- D+M → D → M (Experimental): D : DA-1229 5mg qd, M : metformin 1000mg bid
  Interventions: Drug: DA-1229; Drug: metformin; Drug: DA-1229 + metformin

INTERVENTIONS:
Drug: DA-1229
Drug: metformin
Drug: DA-1229 + metformin

SUMMARY:
This is a randomized, open-label, multiple dosing, three-way crossover clinical trial to investigate the pharmacokinetic/pharmacodynamic drug-drug interaction of DA-1229 5 mg and Metformin IR 1000 mg after oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45, healthy male subjects(at screening)
* Body weight between 55kg - 90kg, BMI between 18.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology, immunology, pulmonary, endocrine, hematooncology, cardiology, mental disorder)
* Subject who had GI tract disease(Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery(appendectomy, hernioplasty are excluded)
* Subject who had drug(Aspirin, antibiotics) hypersensitivity reaction
* Subject who already participated in other trials in 2 months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 months or transfusion in 1 months currently.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of DA-1229 and metformin | up to 168h
Cmax,ss of DA-1229 and metformin | up to 168h

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea